CLINICAL TRIAL: NCT01167244
Title: Phase 2 Trial of BMS-690514 in Non-Small Cell Lung Cancer Subjects Who Have Been Treated With Gefitinib or Erlotinib and Are Genotypically EGFR Mutation Positive or Who Have Had a Prior Response
Brief Title: Trial of BMS-690514 in Non-Small Cell Lung Cancer Subjects Who Have Been Treated With Gefitinib or Erlotinib and Are Genotypically EGFR Mutation Positive or Who Have Had a Prior Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA187-020
Record Dates: First submitted 2010-07-16; First posted 2010-07-22 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — BMS-690514

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-690514 (Experimental)
  Interventions: Drug: BMS-690514

INTERVENTIONS:
Drug: BMS-690514 — Tablets, Oral, 200 mg, once daily, until disease progression or toxicity

SUMMARY:
The purpose of this study is to observe an improvement in overall response rate in NSCLC subjects who have been treated with gefitinib or erlotinib and are genotypically EGFR mutation positive or who have had a prior a response.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent, metastatic or progressive NSCLC without any indication of radiotherapy. Subjects must have:
* Pathologically confirmed NSCLC
* Previously received treatment with single agent Gefitinib or Erlotinib and completed treatment at least 2 weeks prior to study entry
* Any one of the following:
* A tumor that harbors an EGFR mutation
* Objective clinical benefit from treatment with Gefitinib or Erlotinib as defined by either documented and confirmed partial or complete response (RECIST or WHO), or significant and durable (≥ 6 months) clinical benefit (stable disease as defined by RECIST or WHO) Progression of NSCLC while on continuous treatment with gefitinib or erlotinib as noted by CT/MRI increase in disease after having a confirmed partial or complete response or evidence of ≥ 6 months of SD within 3 months of study enrollment

Exclusion Criteria:

* Symptomatic brain metastasis
* History of TIA, CVA, or thrombotic/thromboembolic event (within last 6 months)
* History of hemoptysis greater than 10 mL/day within last 30 days
* Uncontrolled or significant cardiovascular disease
* History of uncontrolled diarrhea, Crohn's disease or ulcerative colitis
* Inability to swallow tablets, untreated malabsorption or GI surgery that results in inability to absorb protocol therapy
* Women unwilling to avoid pregnancy or use adequate contraception
* History of allergy or adverse drug reaction to gefitinib or erlotinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To estimate objective response rate in NSCLC subjects who have been treated with gefitinib or erlotinib and are genotypically EGFR mutation positive or who have had a prior a response | Tumor assessment Day 29 and every 8 weeks from Day 1 thereafter until disease progression
To estimate objective response rate in NSCLC subjects who have been treated with gefitinib or erlotinib and are genotypically EGFR mutation positive or who have had a prior a response | Tumor assesments on Day 29 by CT or MRI
To estimate objective response rate in NSCLC subjects who have been treated with gefitinib or erlotinib and are genotypically EGFR mutation positive or who have had a prior a response | Tumor assessments every 8 weeks from Day 1 by CT or MRI

SECONDARY OUTCOMES:
To estimate disease control rate and progression free survival in all treated subjects | Tumor assessment Day 29 and every 8 weeks from Day 1 thereafter until disease progression
To estimate disease control rate and progression free survival in all treated subjects | Tumor assessment from Day 29
To estimate disease control rate and progression free survival in all treated subjects | Tumor assessment every 8 weeks from Day 1 until disease progression
To evaluate safety and tolerability of BMS-690514 in all treated subjects | Average about 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Japan (4):
  - Local Institution, Kashiwa-Shi, Chiba
  - Local Institution, Osaka-Sayama-Shi, Osaka
  - Local Institution, Sunto-Gun, Shizuoka
  - Local Institution, Koto-Ku, Tokyo

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx